CLINICAL TRIAL: NCT01535209
Title: Phase 3 Study of Stereotactic Radiotherapy of the Postoperative Resection Cavity Versus Whole-Brain Irradiation After Surgical Resection of Single Brain Metastasis
Brief Title: Stereotactic Radiotherapy of Resection Cavity For Single Brain Metastasis Versus Whole-Brain Radiotherapy After Resection
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Maria Sklodowska-Curie National Research Institute of Oncology (Other)
Collaborators: Lower Silesian Oncology Center (Unknown); Copernicus Memorial Hospital (Other); Prof. Franciszek Lukaszczyk Memorial Oncology Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAVITY
Record Dates: First submitted 2012-02-14; First posted 2012-02-17 (Estimated); Last update posted 2012-02-17 (Estimated); Status verified 2012-02

CONDITIONS: Brain Metastases
Keywords: Stereotactic radiotherapy; Whole-brain radiotherapy; Resection cavity
MeSH Terms: conditions — Brain Neoplasms | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SBRT to resection cavity (Experimental): 18Gy in 1 fraction for resection cavity <2cm in maximum diameter, 15Gy in 1 fraction for resection cavity 2.1-3cm in maximum diameter, 15Gy in 1 fraction or 25 Gy in 5 fractions over 5 days for resection cavity 3.1-4cm in maximum diameter, 25 Gy in 5 fractions over 5 days for resection cavity >4cm in maximum diameter
  Interventions: Radiation: stereotactic body radiotherapy (SBRT)
- WBRT (Active Comparator): 30Gy in 10 fractions over 12 days to whole brain
  Interventions: Radiation: Whole-Brain Radiotherapy (WBRT)

INTERVENTIONS:
Radiation: stereotactic body radiotherapy (SBRT) — 18Gy in 1 fraction for resection cavity <2cm in maximum diameter, 15Gy in 1 fraction for resection cavity 2.1-3cm in maximum diameter, 15Gy in 1 fraction or 25 Gy in 5 fractions over 5 days for resection cavity 3.1-4cm in maximum diameter, 25 Gy in 5 fractions over 5 days for resection cavity >4cm in maximum diameter
  Other Names: stereotactic body radiotherapy
  Arms: SBRT to resection cavity
Radiation: Whole-Brain Radiotherapy (WBRT) — 10 x 3 Gy to whole brain
  Other Names: whole brain irradiation; adjuvant cranial irradiation
  Arms: WBRT

SUMMARY:
Adjuvant whole-brain radiation therapy (WBRT) after resection of single brain metastasis is considered as a standard associated with side effects leading to decreased neurocognitive function. The Investigators addressed the question whether stereotactic radiotherapy of the resection cavity impairs neurological status and/or cognitive functions in compare to adjuvant WBRT.

DETAILED DESCRIPTION:
Patients with surgically removed single brain metastasis are randomly allocated to control or experimental arm. Before treatment the MRC Neurological Status Scale is used for assessing neurological status, the EORTC QLQ-C30 and QLQ-BN20 for quality of life and Mini-Mental State Examination to assess cognitive functioning. The control group receive 30Gy in 10 fractions of 3Gy over 12 days to the whole brain. The patients in the experimental arm are treated with stereotactic radiotherapy to the resection cavity. The dose to the tumor bed is 15-18Gy in one fraction or 25Gy in 5 fractions. The study hypothesis is that the difference in the 5-months failure free survival rate isn't higher than 25% in experimental arm compared to control arm.

ELIGIBILITY:
Inclusion Criteria:

* Patients with surgically removed histologically proven metastatic cancer
* Subtotal or total resection of single brain metastasis
* Presence of single brain metastasis in MRI
* Karnofsky Performance Status ≥ 70
* Life expectancy > 6 months (minimal extracranial disease or availability of effective oncology treatment)
* No previous history of cranial irradiation
* Availability of MRI
* Starting radiotherapy within six weeks after neurosurgery
* Negative pregnancy test for woman
* Written informed consent

Exclusion Criteria:

* Dementia and central nervous system diseases leading to higher risk of radiation toxicity
* Contraindications for MRI and/or no patient's tolerance and acceptance of cranial MRI
* Altered level of consciousness
* Histologically proven metastatic small cell lung cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2012-01; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Failure-free survival | 5 months after radiotherapy
  Time to decrease in MRC scale by 1 point or in MMSE by 3 points or neurologic death.

SECONDARY OUTCOMES:
Overall survival | 2 years
Quality of life assessment | 2 years
Time to distant intracranial progression | 2 years
Time to local progression | 2 years
  Time to progression in the irradiated cavity

CONTACTS AND LOCATIONS:
Overall Officials: Lucyna Kepka, Prof., Principal Investigator — M.Sklodowska-Curie Memorial Cancer Centre, Warsaw, Poland
Locations (1):
- M.Sklodowska-Curie Memorial Cancer Centre, Warsaw, Poland